CLINICAL TRIAL: NCT00713310
Title: Study to Assess the Safety and Efficacy of Asacol® (1.2 to 4.8 g/Day) Administered as 400 mg Delayed-release Tablets Given Every 12 Hours for 6 Weeks to Children and Adolescents With Mildly-to-Moderately Active Ulcerative Colitis
Brief Title: Assessing the Safety/Efficacy of Asacol® Given Every 12 Hours to Children and Adolescents With Active Ulcerative Colitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Warner Chilcott (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2007017
Record Dates: First submitted 2008-07-09; First posted 2008-07-11 (Estimated); Results first posted 2012-04-04 (Estimated); Last update posted 2012-04-05 (Estimated); Status verified 2012-04

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Mesalamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Low-Dose (Experimental): 1.2 - 2.4 g/day Asacol dependent on body weight
  Interventions: Drug: Asacol 400 mg
- High-Dose (Experimental): 2.0 - 4.8 g/day Asacol dependent on body weight
  Interventions: Drug: Asacol 400 mg

INTERVENTIONS:
Drug: Asacol 400 mg — High dose:
  17-<33 kg = 3 Asacol 400mg in morning and 2 Asacol 400 in PM, 33-<54 kg = 5 Asacol 400mg in morning and 4 Asacol 400 in PM, 54-<90 kg = 6 Asacol 400mg in morning and 6 Asacol 400 in PM
  Arms: High-Dose
Drug: Asacol 400 mg — Low dose:
  17-<33 kg = 2 Asacol 400mg + 1 placebo in morning and 1 Asacol 400 +1 placebo in PM, 33-<54 kg = 3 Asacol 400mg +2 placebo in morning and 2 Asacol 400 + 2 placebo in PM, 54-<90 kg = 3 Asacol 400mg + 3 placebo in morning and 3 Asacol 400mg + 3 placebo in PM
  Arms: Low-Dose

SUMMARY:
The overall objective of this study is to assess the safety and efficacy of high dose and low dose Asacol administered as 400 mg delayed-release tablets given every 12 hours for 6 weeks to children and adolescents with mildly-to-moderately active ulcerative colitis.

ELIGIBILITY:
Inclusion Criteria:

* are male or female between the ages of 5 and 17 years, inclusive, at the time of the first dose of study medication, with a history of biopsy and endoscopy confirmed UC;
* have mildly-to-moderately active UC (either newly diagnosed or that has relapsed) as defined clinically by a Pediatric UC Activity Index (PUCAI) score 10 and 55, and, in the opinion of the Investigator, the patient does not require steroids;
* have baseline scores of at least 1 for both rectal bleeding (Streaks of blood with stool less than half of the time) and stool frequency (1-2 stools greater than normal per day) as defined by the TM-Mayo Score

Exclusion Criteria:

* have UC known to be confined to the rectum (isolated rectal proctitis);
* have a history of allergy or hypersensitivity to salicylates, aminosalicylates, or any component of the Asacol tablet;
* have a significant co-existing illness or other condition(s), including but not limited to cancer or significant organic or psychiatric disease on medical history or physical examination, that, in the judgment of the Investigator, contraindicate(s) administration of the study drug and/or any study procedures

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 83 (Actual)
Dates: Start 2008-12; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Preston M Dunnmon, MD, Study Director — Procter and Gamble
Locations (40):
- United States (25):
  - Research Facility, Birmingham, Alabama
  - Research Facility, Phoenix, Arizona
  - Research Facility, Loma Linda, California
  - Research Facility, San Diego, California
  - Research Facility, San Francisco, California
  - Research Facility, Washington D.C., District of Columbia
  - Research Facility, Gainesville, Florida
  - Research Facility, Park Ridge, Illinois
  - Research Facility, Louisville, Kentucky
  - Research Facility, Boston, Massachusetts
  - Research Facility, Worcester, Massachusetts
  - Research Facility, Kansas City, Missouri
  - Research Facility, Omaha, Nebraska
  - Research Facility, Mays Landing, New Jersey
  - Research Facility, Buffalo, New York
  - Research Facility, New Hyde Park, New York
  - Research Facility, Youngstown, Ohio
  - Research Facility, Portland, Oregon
  - Research Facility, Chattanooga, Tennessee
  - Research Facility, Knoxville, Tennessee
  - Research Facility, Fort Worth, Texas
  - Research Facility, Houston, Texas
  - Research Facility, San Antonio, Texas
  - Research Facility, Norfolk, Virginia
  - Research Facility, Huntington, West Virginia
- Canada (5):
  - Research Facility, Halifax, Nova Scotia
  - Research Facility, Hamilton, Ontario
  - Research Facility, London, Ontario
  - Research Facility, Ottawa, Ontario
  - Research Facility, Montreal, Quebec
- Croatia (2):
  - Research Site, Rijeka, Croatia
  - Research Site, Zagreb, Croatia
- Poland (6):
  - Research Site, Bialystok, Poland
  - Research Site, Bydgoszcz, Poland
  - Research Site, Krakow, Poland
  - Research Site, Lodz, Poland
  - Research Site, Warsazawa, Poland
  - Research Site, Wroclaw, Poland
- Romania (2):
  - Research Site, Bucharest, Romania
  - Research Site, Iași, Romania

REFERENCES:
- [Derived] Winter HS, Krzeski P, Heyman MB, Ibarguen-Secchia E, Iwanczak B, Kaczmarski M, Kierkus J, Kolacek S, Osuntokun B, Quiros JA, Shah M, Yacyshyn B, Dunnmon PM. High- and low-dose oral delayed-release mesalamine in children with mild-to-moderately active ulcerative colitis. J Pediatr Gastroenterol Nutr. 2014 Dec;59(6):767-72. doi: 10.1097/MPG.0000000000000530. PMID 25419597

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment began 16 Dec 2008
Groups:
- Low-Dose: 17-<33kg: AM - 2 Asacol 400mg & 1 placebo, PM - 1 Asacol 400mg & 1 placebo; 33-<54kg: AM - 3 Asacol 400mg & 2 placebo, PM - 2 Asacol 400mg & 2 placebo; 54-<90kg: AM & PM - 3 Asacol 400mg & 3 placebo
- High-Dose: 17-<33kg: AM 3 Asacol 400mg, PM 2 Asacol 400mg; 33-<54kg: AM5 Asacol 400mg, PM 4 Asacol 400mg; 54-<90kg: AM & PM 6 Asacol 400mg
Period: Overall Study
Arm/Group | Low-Dose | High-Dose
Started | 41 | 42
mITT Population | 41 | 41 (1 subject randomized to high dose not dosed so not included in the mITT population.)
Completed | 36 | 36
Not Completed | 5 | 6
Not completed — Adverse Event | 5 | 2
Not completed — Lack of Efficacy | 0 | 2
Not completed — Withdrawal by Subject | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Low-Dose | High-Dose | Total
Number analyzed (Participants) | 41 | 42 | 83
Age Continuous [Mean (Standard Deviation); unit: years] — mITT Population
  years | 13.0 (3.2) | 12.8 (3.0) | 12.9 (3.1)
Age, Customized [Number; unit: participants]
  5-8 years | 4 | 4 | 8
  9-17 years | 37 | 38 | 75
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 23 | 45
  Male | 19 | 19 | 38
Region of Enrollment [Number; unit: participants]
  United States | 26 | 23 | 49
  Canada | 0 | 4 | 4
  Poland | 9 | 10 | 19
  Romania | 2 | 3 | 5
  Croatia | 4 | 2 | 6

OUTCOME MEASURES:

1. Primary Outcome: Treatment Success PUCAI (Pediatric Ulcerative Colitis Activity Index), mITT/Modified Intent to Treat Population
Description: PUCAI 0-85, abdominal pain (no pain/0, pain ignored/5, pain not ignored/10), rectal bleeding (none/0, small <50% stool/10, small with most stools/20, large >50% stool/30), stool consistency (formed/0, partially/5, unformed/10), # per 24 hrs (0-2/0, 3-5/5, 6-8/10, >8/15), nocturnal bowel movements (no/0, yes/10), activity level (no limitation/0, occasional limitation/5, severely restricted/10) Remission <10, Mild 10-34, Moderate 35-64, Severe 65-85, Success score<10 at Wk 6 (complete) or reduction of >=20 points baseline to Wk 6 with Wk 6 score>=10 (partial)
Time Frame: Baseline and 6 weeks
Population: miTT includes subjects who were randomized and took at least one dose of study medication
Measure: Number; unit: % participants with treatment success
Groups:
- Low Dose: Low Dose = Asacol 1.2 - 2.4 g/day stratified based on weight (17-<33 kg, 33-<54 kg, 54-90 kg) & disease severity (mild/moderate)
- High Dose: High Dose = Asacol 2.0 - 4.8 g/day based on weight (17-<33 kg, 33-<54 kg, 54-90 kg) & disease severity (mild/moderate)
Arm/Group | Low Dose | High Dose
Number analyzed (Participants) | 41 | 41
% participants with treatment success | 56.1 | 55.0
Statistical Analysis 1: Comparison: Low Dose vs High Dose; A total of about 100 subjects were to be enrolled in the study with the expectation that about 80 subjects (40/dose level) would complete. Minimum of 9 subjects in 5-8 year old range were to be enrolled, 4-5 per dose level (high/low). A 2-sided α=0.05 Fisher's Exact test has an estimated power of P=0.50 with 40 subjects per dose level; Test type: Superiority or Other; p = 0.9240, Cochran-Mantel-Haenszel; High-Low Dose Difference Success Rates = -1.1, 95% CI 2-sided [-22.7 to 20.5]

2. Secondary Outcome: Treatment Success PUCAI Amended Endpoint (5 Point Scale Abdominal Pain), mITT
Description: PUCAI 0-85, abdominal pain amended (no pain/0, very mild/2.5, mild/5, moderate/7.5, severe/10), rectal bleeding (none/0, small <50% stool/10, small with most stools/20, large >50% stool/30), stool consistency (formed/0, partially/5, unformed/10), # per 24 hrs (0-2/0, 3-5/5, 6-8/10, >8/15), nocturnal bowel movements (no/0, yes/10), activity level (no limitation/0, occasional limitation/5, severely restricted/10) Remission <10, Mild 10-34, Moderate 35-64, Severe 65-85, Success score<10 at Wk 6 (complete) or reduction of >=20 points baseline to Wk 6 with Wk 6 score>=10 (partial)
Time Frame: Baseline and Week 6
Population: mITT subjects who were randomized & took at least one dose of study medication
Measure: Number; unit: % participants with treatment success
Arm/Group | Low Dose | High Dose
Number analyzed (Participants) | 41 | 41
% participants with treatment success | 56.1 | 57.5
Statistical Analysis 1: Comparison: Low Dose vs High Dose; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.8193, Cochran-Mantel-Haenszel; High-Low Dose Difference Success Rates = 1.4, 95% CI 2-sided [-20.2 to 23.0]

ADVERSE EVENTS:
Time Frame: Day -7 thru Week 6 of trial (7 weeks)
Arm/Group | Low Dose | High Dose
Serious Adverse Events (participants affected / at risk) | 5/41 | 2/41
Other Adverse Events (participants affected / at risk) | 20/50 | 15/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Low Dose (N=41) | High Dose (N=41)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Body Mass Index Decreased (Investigations) | 1 (1) | 0 (0)
Colitis Ulcerative (Gastrointestinal disorders) | 1 (1) | 1 (1)
Adenovirus Infection (Infections and infestations) | 1 (1) | 0 (0)
Diarrhoea Haemorrhagic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Cholangitis Sclerosing (Hepatobiliary disorders) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Low Dose (N=50) | High Dose (N=41)
Colitis Ulcerative (Gastrointestinal disorders) | 5 (5) | 2 (2)
Fatigue (General disorders) | 1 (1) | 3 (3)
Pyrexia (General disorders) | 0 (0) | 3 (3)
Nasopharyngitis (Infections and infestations) | 4 (4) | 4 (4)
Sinusitis (Infections and infestations) | 3 (3) | 0 (0)
Dizziness (Nervous system disorders) | 3 (3) | 1 (1)
Headache (Nervous system disorders) | 4 (4) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less